CLINICAL TRIAL: NCT06312410
Title: The VIA Family 2.0 Study: a Randomized Clinical Trial Evaluating Family-based Interventions for Children Born to Parents with Mental Disorders
Brief Title: The VIA Family 2.0 - a Family Based Intervention for Families with Parental Mental Illness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Aalborg Psychiatric Hospital (Other); TrygFonden, Denmark (Industry); Novo Nordisk A/S (Industry); Lundbeck Foundation (Other); Liljeborgfonden (Unknown); Ebbefos Fonden (Unknown); KV Fonden (Unknown)
Responsible Party: Principal Investigator, Anne Amalie Elgaard Thorup, Clinical professor, PhD, MD, specialist in child and adolescent psychiatry, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-23067714
Record Dates: First submitted 2024-02-28; First posted 2024-03-15 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-03

CONDITIONS: Child; Parents; Mental Disorder; Child of Impaired Parents; Preventive Health Services
Keywords: family based intervention; early intervention; familial high risk; COPMI - children of parents with mental illness; parental mental illness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VIA Family 2.0 (Experimental): In the intervention all child-involving elements are adapted to the specific age groups of the children, but everything is built on the same basic multidisciplinary, holistic and cross-sectional team model.
  Every family will be affiliated to a case manager, who will coordinate all activities and appointments and be available throughout the intervention period of two years. A range of intervention elements will be offered to the family, depending on age of the child(ren), the family's needs and will always rely on their motivation:
  * Case-management supporting to reach good family functioning
  * Family-based psychoeducation
  * Parents' and children's groups with integrated peer-support
  * Parenting support and training
  * Mapping and nurturing of resources in the social network and social counseling
  * Early assessment of children's possible mental health problems
  * All elements will be adapted to the age of the children (details available upon request)
  Interventions: Other: VIA Family 2.0
- Treatment as usual (TAU) (Active Comparator): TAU varies to some extent in the two regions, but common is that it consists of 2-3 family consultations (family sessions) with the presence of parents and all children above the age of six years.
  These consultations will be managed by the Center for Relatives in the North Denmark Region and by the clinical 'child key persons' , who are staff with a special training in children and family impact in all departments of mental health services in the Capital Region.
  The child is also referred to participate in a psychoeducational group for same aged children. Children can participate in a group with peers, who have a parent with a mental illness as well. These groups are run by two therapists with many years of experience working with groups like this for different age groups. Participation in groups like this is voluntary, and not all children continue in a group after the family consultations.
  Interventions: Other: VIA Family 2.0

INTERVENTIONS:
Other: VIA Family 2.0 — Multidisciplinary team based preventive intervention. For details, please see arm/group description.

SUMMARY:
VIA Family 2.0 - a Family Based Intervention for families with parental mental illness

Background: Children born to parents with mental illness have consistently been shown to have increased risks for a range of negative life outcomes including increased frequencies of mental disorders, somatic disorders, poorer cognitive functioning, social, emotional and behavioral problems and lower quality of life. Further these children are often overlooked by both society and mental health services, although they represent a potential for prevention and early intervention.

A collaboration between researchers and clinicians from two regions, the Capital Region and the North Region Denmark has been established as the Research Center for Family Based Interventions. The research center is an umbrella for a series of research activities, all focusing on children and adolescents in families with parental mental illness.

Method: A large randomized, controlled trial (RCT) for families with parental mental illness will be conducted in order to evaluate the effect of a two-year multidisciplinary, holistic team intervention (the VIA Family 2.0 team intervention) against treatment as usual (TAU). Inclusion criteria will be biological children 0-17 of parents with any mental disorder treated in the secondary sector at any time of their life and receiving treatment in primary or secondary sector within the previous three years. A total of 870 children or approx. 600 families will be included from two sites. Primary outcomes will be changes in child well being, parental stress, family functioning and quality of the home environment, .

Time plan: The RCT will start including families from March 1st, 2024 to Dec 2025 (or later if needed). All families will be assessed at baseline and at end of treatment, i.e. after 24 months and after 36 months. Baseline data will inform the intervention team about each family's needs, problems, and motivation. TAU will be similar in the two regions, which means three family meetings and option for children to participate in peer groups.

Challenges: final funding is being applied for. Recruitment of families can be challenging but we have decades of experience in conducting research in the field. Since both the target group, their potential problems and the intervention is complex, primary outcome is difficult to determine.

DETAILED DESCRIPTION:
A detailed study protocol will be published in 2024

ELIGIBILITY:
Inclusion Criteria:

* At least one of the parents must be living in Capital Region or in Region North, Denmark, and at least one biological child under age 18 must be living with one of the parents. Only biological children of the parent with at mental health problem can be included.
* The parent with the mental health problems has at some point been diagnosed in the secondary sector and has within the last three years been treated in the primary sector (GP or private psychiatric clinic) or in the secondary sector (hospital psychiatry).
* Patients with substance abuse can only be included if substance abuse is a secondary diagnosis to another mental illness disorder being treated within the secondary sector during the last three years.
* All adult participants must give informed consent. Both parents will need to consent in case of shared custody, but do not have to participate if they are reluctant to do so.

Exclusion Criteria:

* Not fulfilling inclusion criteria
* Not giving informed consent
* Living at Læsø or at Bornholm, Denmark
* Children placed in care outside of the home fulltime in institution of professional family care (the family is not excluded if the children placed in part time in care outside home or fulltime family care within the family)
* No risk factors found after baseline assessment (as described in the stepped care model) at baseline - these families can be re-referred if their situation changes.
* Ongoing intensive family treatment in the municipality (for example staying at an institution for parental evaluation by the authorities)?

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1452 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Strengths and Difficulties Questionnaire (SDQ) | Baseline, end of intervention (24 months) and 36 months follow up.
  Primary outcome for children/adolescents aged 3 years to 17 years will be child's development and wellbeing measured by Strengths and Difficulties Questionnaire (SDQ), which has been used in several other studies, is easy to complete, has Danish norms and is a part of the diagnostic evaluation, Development and Well-Being Assessment, (DAWBA), will be used for psychopathology assessment as well, and can be filled in digitally by the primary caregiver before the clinical assessment. The higher score, the more problems Rated by child from age 11 and by always by parent. A 25 item self-report questionnaire assessing developmental, behavioural and emotional problems completed by children aged 11-17. Items are rated on a three-point Likert scale (0= not true, 1= somewhat true, 2= certainly true).
Change in Bayley-4 Bayley Scales Test for Infant and Toddler Development | Baseline, after 6 months, after 12 months, after 18 months and after 24 months.
  The primary outcome for the youngest children aged 0-2 years will be scores from Bayley-4, a clinical test of the child's cognitive, language, motor and emotional development, conducted by a trained researcher. Scores range from 1-19, the higher score the better functioning
Change in Family Assessment Device - General Function Scale (FAD-GF) | Baseline, end of intervention (24 months), and 36 months follow up
  Primary outcome for the whole family is family functioning rated by the primary caregiver. Family function will be measured by the questionnaire Family Assessment Device, a 12 item questionnaire by the parents and children from age 12 Scale from 1-4. Low score represents better outcome.
Change in Parental Stress Scale (PSS) | Baseline, end of intervention (24 months) and 36 months follow up.
  The primary outcome for the parents is parental stress measured by the Parental Stress Scale (PSS), which is a 18 item parent-reported questionnaire on the quality of experienced stress related to parenting. Score 1-5. A higher score indicates more parental stress.

SECONDARY OUTCOMES:
Change in Home Observation for Measurement of the Environment (HOME) | Baseline, end of intervention (24 months) and 36 months follow up.
  A clinician rated semi-structured interview with both caregiver and child measuring stimulation and support in the home environment (scale 0-60/62 dep on age versions). Higher score represents better outcome.
Change in Parenting and Family Adjustment Scales (PAFAS) | Baseline, end of intervention (24 months), and 36 months follow up
  30 item questionnaire assessing changes in parenting practices, parental adjustment, and family relationships. Scores from 0-90, higher scores indicates poorer parenting or adaptation
Change in Children's Global Assessment Scale (CGAS) | Baseline, end of intervention (24 months) and 36 months follow up
  A clinical rated measurement based on interview to assess general functioning in children. Information is obtained from the child and the caregiver, separately. Scale from 1-100. Higher score indicates better functioning.
Change in Perceived Stress Scale (PSS) | Baseline, end of intervention (24 months) and 36 months follow up.
  10 item questionnaire measuring perceived stress (parents)
Client Satisfaction Scale (CSQ) | End of intervention (24 months)
  Questionnaire with 8 items measuring patient/client .Total scores range from 8 to 32, with the higher number indicating greater satisfaction.

OTHER OUTCOMES:
Change in Ages and Stages Questionnaire:SE-2 (ASQ-SE) | Baseline, after 6 months, after 12 months, after 18 months, after 24 months and 36 months (for children aged 3-5 years)
  Questionnaire measuring child social and emotional development and milestones. Scores range from 0-465, higher scores above cut-off (59) indicate social and emotional problems.
Change in Daily Life Stressor Scale (DLSS) | Baseline, end of intervention (24 months) and 36 months follow up.
  14 item questionnaire measuring child stress, scores range from 0-56, the higher score the higher level of perceived stress
Change in Child and Youth Resilience Measure (CYRM-R) | Baseline, end of intervention (24 months) and 36 months follow up.
  A 12 item self-report questionnaire from age 5 assessing resiliency in children across a number of areas including personal skills, peer support, social skills, physical and psychological caregiving, educational and cultural. Items are rated on a 3- or 5-point Likert scale. Higher scores indicating greater resiliency.
Alarm Distress Baby Scale (ADBB) | Baseline, after 6 month (for children age 0-2 years), after 12 month, after 18 months, after 24 months), and 36 months follow up
  Test for children aged 2-24 months measuring social withdrawal, scores range from 0-32, scores above 4 indicate social withdrawal, the higher score the more severe
Change in Personal and Social Performance Scale (PSP) | Baseline, end of intervention (24 months) and 36 months follow up.
  An interviewer-rated scale assessing the parent's personal and social functioning over four domains (social activities, social relationships, self-care and aggressive behavior).
  Scores range from 1-100, the higher score the better social functioning.
Change in Warwick Edinburgh Mental Wellbeing Scale (WEMWBS) | Baseline, end of intervention (24 months) and 36 months follow up.
  14 item questionnaire measuring mental wellbeing (non-index parent) scores range from 14 to 70, the higher scores, the better mental wellbeing
Change in Global Assessment of Function - Symptoms (GAF-S) | Baseline, end of intervention (24 months) and 36 months follow up.
  An interviewer-rated scale assessing the Parents Level of Psychiatric Symptoms. GAF-S provides a score from 1-100, with higher scores indicating better outcome.
Change in Kessler Psychological Distress Scale, K10 | Baseline, end of intervention (24 months) and 36 months follow up.
  10 item questionnaire on psychological distress with a five-level response scale. Scale from 10-50. Higher score indicating higher level of psychological distress.
Change in General Self-Efficacy Scale (GSE) | Baseline, end of intervention (24 months) and 36 months follow up.
  10 item questionnaire measuring general belief in one's own capabilities. Self-report. Total score is measured. Ranges from 10 to 40. Higher scores indicates better self-efficacy.
Change in Social Provision Scale-short form (SPS) | Baseline, end of intervention (24 months), and 36 months follow up
  The perceived social network can be understood as a resource for resilience and will be measured with Social Provision Scale (SPS) short form, a.10 item questionnaire, with scores ranging from 10-40, the higher score the better social provision perceived
Change in Quality-adjusted life year (EQ-5D) | Baseline, end of intervention (24 months) and 36 months follow up.
  6 item questionnaire, range from 0-100, the higher score the better health
Change in Self-Stigma of Mental Illness Scale - short form (SSMIS-SF) | Baseline, end of intervention (24 months) and 36 months follow up.
  20 item questionnaire on mental health self-stigma (only index parent), in four subscales (stereotype awareness, stereotype agreement, application to self , harm to self-esteem), each scoring from 5 (low) to 45 (high).
Change in The Questionnaire about the Process of Recovery (QPR) | Baseline, end of intervention (24 months) and 36 months follow up.
  15 item questionnaire on the process of recovery on a 4-point scale. Higher scores are indicative of recovery. Only index parent.
General Intelligence Test (RIST) | Baseline
  A clinician rated test measuring general intelligence. The RIST comprises a verbal subtest (Guess What) and a nonverbal subtest (Odd-Item Out).
  Guess What is a classic measure of crystallized intelligence, whereas Odd-Item Out shares characteristics with fluid intelligence.

CONTACTS AND LOCATIONS:
Locations (1):
- VIA Family 2.0 at BFOR, Gentofte Hospitalsvej 3A, Gentofte Hospital, Copenhagen, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No